CLINICAL TRIAL: NCT03589560
Title: Clinical and Radiographic Evaluation of Biodentine and Mineral Trioxide Aggregate in Revascularization of Non Vital Immature Permanent Anterior Teeth (Randomized Clinical Study)
Brief Title: Evaluation of Biodentine and Mineral Trioxide Aggregate in Revascularization of Non Vital Immature Anterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Mohsen Aly, Assistant Lecturer of Pediatric Dentistry and Dental public health, Faculty of Dentistry, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pulp revascularization
Record Dates: First submitted 2018-06-24; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Pulp Necrosis
Keywords: revascularization; necrotic; immature; coronal plug
MeSH Terms: conditions — Dental Pulp Necrosis; Necrosis | interventions — tricalcium silicate; mineral trioxide aggregate; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine (Experimental): 3-4 mm of Biodentine (Septodont, St. Maur-des-Fosses, France) was applied over the clot carefully in group I by using amalgam carrier. material was packed lightly with a moistened cotton pellet and Periapical radiograph was taken to confirm coronal seal in the second visit of dental pulp revascularization.
  Interventions: Drug: Biodentine
- Mineral Trioxide Aggregate (Active Comparator): 3-4 mm of white Mineral Trioxide Aggregate (Angelus, Londrina, Brazil) was applied over the clot in group II by using amalgam carrier. material was packed lightly with a moistened cotton pellet and Periapical radiograph was taken to confirm coronal seal in the second visit of dental pulp revascularization.
  Interventions: Drug: Mineral Trioxide Aggregate

INTERVENTIONS:
Drug: Biodentine — a procedure used to regenerate a pulp-dentine complex that restores functional properties of this tissue, fosters continued root development for immature teeth, and prevents or resolves apical periodontitis.
  Other Names: Dentine substitute material
  Arms: Biodentine
Drug: Mineral Trioxide Aggregate — a procedure used to regenerate a pulp-dentine complex that restores functional properties of this tissue, fosters continued root development for immature teeth, and prevents or resolves apical periodontitis.
  Other Names: MTA
  Arms: Mineral Trioxide Aggregate

SUMMARY:
the object of this study is to evaluate clinically and radiographically the effect of using Biodentine and Mineral Trioxide Aggregate as coronal plug materials in revascularization of non-vital immature teeth

DETAILED DESCRIPTION:
Traumatic injury to the anterior teeth is commonly found among young children, represent one third in boys and one fourth in girls. Because the root development completed two years after eruption of the tooth into the oral cavity, an incomplete root development is one of the most common complication seen in traumatized teeth. Loss of pulp vitality before dentine deposition is completed, leaves a weak root more susceptible to fracture as a result of the thin dentinal walls. It will also lead to a poor crown/root ratio, with possible periodontal injury as a result of increased mobility.

Several techniques have been advocated to manage the open apex of immature teeth, including calcium hydroxide (Ca(OH)2) apexification or apical barrier technique with Mineral Trioxide Aggregate (MTA). Although these techniques were successful in obtaining apical closure and healing of the apical pathosis, they have certain disadvantages, as the root walls of the immature tooth remain thin and short as hard tissue barrier formation only occurs apically, with no further root development.

As an replacement to traditional methods, the use of a regenerative endodontic procedure has been recommended as it may strengthen the root walls through the deposition of hard tissue and promote the development of a normal apical morphology. MTA was chosen to be placed over blood clot to provide excellent seal and it was considered the recommended material for regenerative procedures.The application of MTA over a blood clot was technically difficult, and condensation resulted in displacement of the material apically. Another important note was the prolonged setting time of MTA which resulted in postponing placement of composite restoration to next appointments and post-treatment tooth discoloration.

Biodentine has the same mechanical properties as human dentine, very low cytotoxicity and overcome clinical drawbacks of white MTA. It had better consistency and allow its condensation without any apical displacement. Biodentine sets within twelve minutes, which allow placement of composite restoration in the same appointment. Biodentine is tooth-colored and doesn't cause the discoloration resulted from the presence of the material at level of the orifice.

ELIGIBILITY:
Inclusion Criteria:

* Patients free from any systemic diseases that may hinder the normal healing process.
* Age from 8-15 y
* Tooth with immature root apex (apical opening greater than 1mm)
* Traumatically or cariously exposed single rooted teeth
* Non vital permanent anterior tooth with apical periodontitis/abscess
* Pulp space not requiring post and core for final restoration.

Exclusion Criteria:

* Patients having allergy to medicaments or antibiotics necessary to complete procedure.
* Tooth with vital pulp or complete root formation.
* Teeth with internal or external root resorption.
* Un-cooperative patient

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
pain on biting | 3 months
  Binary outcome (Present or absent). Assessed by asking the patient
pain on biting | 6 months
  Binary outcome (Present or absent). Assessed by asking the patient
pain on biting | 9 months
  Binary outcome (Present or absent). Assessed by asking the patient
pain on biting | 12 months
  Binary outcome (Present or absent). Assessed by asking the patient

SECONDARY OUTCOMES:
pain on percussion | 3, 6, 9, 12 month
  Binary outcome (Present or absent). Assessed by tapping the tooth with the back of the mirror
swelling | 3, 6, 9, 12 month
  Binary outcome (Present or absent). Assessed by visual examination of labial vestibule
mobility | 3, 6, 9, 12 month
  Binary outcome (Present or absent). Assessed by applying pressure with the ends of 2 metal instruments
Sinus or fistula | 3, 6, 9, 12 month
  Binary outcome (Present or absent). Assessed by visual examination of labial vestibule
crown discoloration | 3, 6, 9, 12 month
  Binary outcome (Present or absent). Assessed by visual examination of the crown
root lengthening | 3, 6, 9, 12 month
  Evaluated radiographically using DIGORA software.Unit of measurements were mm
root lengthening | 3, 6, 9, 12 month
  Evaluated radiographically using DIGORA software.Unit of measurements were percent

CONTACTS AND LOCATIONS:
Overall Officials: Randa Youssef, PHD, Study Director — Cairo University